CLINICAL TRIAL: NCT05890937
Title: Effect of Mental Stress on Balance in Healthy Adults
Brief Title: Mental Stress on Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Mohammed Torad, Lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P.T/BAS/4/2023/48
Record Dates: First submitted 2023-05-15; First posted 2023-06-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Mental Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mental stress group (Experimental): they were expected to take their exams just after the assessment and before measuring for the second time
  Interventions: Diagnostic Test: Oral and practical exam
- Control group (No Intervention): they were expected to take nothing for 30 min just after the assessment and before measuring for the second time

INTERVENTIONS:
Diagnostic Test: Oral and practical exam — Oral and practical exam that performed at the end of the semester
  Arms: Mental stress group

SUMMARY:
Objectives:

This study aimed to examine the impact of mental stress on balance systems in healthy adults.

Study population & Sample size:

Participants were delimited to 178 students that enter oral and practical exams at different levels in Faculty of Physical Therapy, KafrEl-Sheikh University. Balance was measured using mini-SITCIB test before and after the exam. another 40 subject that have no exam were recruited to work as control group

Study Design :

it is a controlled trial.

Methods :

After obtaining the consent form, and demographics. The mobile application was opened, and a new experiment was created. Abdominal support was modified so it contains a pocket in its centre so the mobile can fit onto it. Participants were asked to conduct a mini-SITCIB test before and after the exam in experimental group and before and after 30 min in control group. The data was extracted and stored anonymously on the hard drive as CSV files.

DETAILED DESCRIPTION:
Mental health is a critical but often overlooked aspect of overall health. Research has shown that mental stress can have detrimental effects on physical health, including balance impairments, in healthy adults. Balance is a crucial physiological function that impacts daily activities and quality of life. Imbalance due to mental stress can increase the risk of falls, injuries, and other health issues, particularly in the aging population.

Objectives:

This study aimed to examine the impact of mental stress on balance systems in healthy adults.

Study population & Sample size:

Participants were delimited to 178 students that enter oral and practical exams at different levels in Faculty of Physical Therapy, KafrEl-Sheikh University. Balance was measured using mini-SITCIB test before and after the exam. another 40 subject that have no exam were recruited to work as control group

Study Design :

it is a controlled trial.

Methods :

After obtaining the consent form, and demographics. The mobile application was opened, and a new experiment was created. Abdominal support was modified so it contains a pocket in its centre so the mobile can fit onto it. Participants were asked to conduct a mini-SITCIB test before and after the exam in experimental group and before and after 30 min in control group. The data was extracted and stored anonymously on the hard drive as CSV files.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 30
* free of any diseases

Exclusion Criteria:

* any trauma within last 2 weeks

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Jerk in X,Y,Z | 2 weeks
  Captured by accelerometer readings
Swaying in X,Y,Z | 2 weeks
  Captured by Gyroscope readings

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh university, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No